CLINICAL TRIAL: NCT05162989
Title: iCare HOME2 Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icare Finland Oy (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TA023-207
Record Dates: First submitted 2021-12-16; First posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Intraocular Pressure; Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Masking Description: Investigator cannot see both the test device and reference device measurement results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- iCare HOME2 vs iCare IC200 (Experimental): Measurement of intraocular pressure (IOP) with iCare IC200 reference tonometer compared to iCare HOME2 test tonometer. Measurement will be performed to categorize each subject as having Low IOP (7 to 16 mmHg), Medium IOP (>16 to <23 mmHg), or High IOP (≥23 mmHg).
  Interventions: Device: iCare HOME2 vs iCare IC200

INTERVENTIONS:
Device: iCare HOME2 vs iCare IC200 — Measurement of IOP with iCare HOME2 compared with iCare IC200.

SUMMARY:
The aim of this clinical study is to provide information about the variability of the intraocular pressure (IOP) self-measurements with the iCare HOME2 tonometer in comparison to the variability of the IOP measurements with the reference tonometer (iCare IC200), over a wide range of IOP values.

DETAILED DESCRIPTION:
The clinical study is planned to estimate the variability of the IOP measurement of iCare HOME2 and IC200. In the study, the subjects will learn to operate the iCare HOME2 tonometer independently by using the labeling materials provided to them. Once they learn to operate the tonometer, subjects will take three self-measurements on the selected eye both in sitting and supine position.

The variability of the measurement results taken with iCare HOME2 will be compared to the variability of the measurement results taken with iCare IC200 by using the recorded results from the study subjects.

ELIGIBILITY:
Inclusion Criteria:

* Glaucoma patients having confirmed optic nerve damage with visual field defects consistent with the glaucomatous optic neuropathy or
* Glaucoma-suspects being followed because of elevated IOP, and/or because of other risk factors for developing glaucoma or optic nerve damage.

Exclusion Criteria:

* Active ocular infection (e.g., pink eye or infectious conjunctivitis)
* Recent trauma to the eye including corneal laceration or corneal/scleral perforation
* Disabling arthritis or difficulty handling the tonometer
* Severe difficulty in opening the eyes including abnormal contractions or twitches of the eyelid (blepharospasm)
* Involuntary, rapid, and repetitive eye movements (nystagmus)
* Low uncorrected near visual acuity of 20/200 or below
* Significant glaucomatous central field loss
* Only one functional eye
* Poor or off-center visual fixation
* Poor hearing and/or communicates using sign language
* Keratoconus (or other corneal disorder)
* Congenitally small eye (microphthalmos)
* Enlarged eyeball from the childhood glaucoma (buphthalmos)
* Previous experience using or interacting with the HOME tonometer during usability tests or clinical trials
* Any affiliation with Icare and its employees
* High corneal astigmatism (>3d)
* History of prior invasive corneal surgery including corneal laser surgery less than six months ago (e.g., LASIK, LASEK, Smile)
* Corneal scarring
* Very thick or very thin corneas (central corneal thickness greater than 600 μm or less than 500 μm)
* Cataract extraction within the last 2 months
* Wearing contact lenses during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-11-26 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Repeatability of IOP measurements | Through study completion, an average of 1-2 months
  Repeatability of IOP measurements comparison of iCare HOME2 vs iCare IC200

CONTACTS AND LOCATIONS:
Overall Officials: Michelle A Sato, MD, Principal Investigator — East West Eye Institute
Locations (1):
- East West Eye Institute, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No